CLINICAL TRIAL: NCT04347577
Title: Investigation Into the Diversity and Dynamic Succession of Gut Flora Pre- and Post-remission in Major Depressive Disorder
Brief Title: Intestinal Flora and Major Depressive Disorders
Acronym: IFMDD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Collaborators: Capital Medical University (Other)
Responsible Party: Principal Investigator, Hui Shi, deputy director, Beijing Chao Yang Hospital
Other Study IDs: HShi
Record Dates: First submitted 2020-04-11; First posted 2020-04-15 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Major Depressive Disorder
Keywords: major depressive disorder; Intestinal flora; remission
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: duloxetine — open-label study
  Other Names: cymbalta

SUMMARY:
As an important micro-ecological factor in human body, intestinal flora is closely related to the occurrence and development of major depressive disorder. The purpose of our study is to investigate a microbiome probe of depression. This study is a 6-months open trial that will enroll approximately 30 patients in major depressive disorders and 10 age- and sex-matched healthy controls. We will comparing gut bacteria community structures of pre- treatment, those of 1 month and 6 months after treatment to remission. With the microbiome change in a preliminary analysis of pre-and post-treatment, we will reveal the diversity before and after the depression treatment.

DETAILED DESCRIPTION:
Participants (30 patients and 10 controls) will be recruited in the clinical psychological department of Beijing Chaoyang hospital. Patients with first-episode major depressive disorder confirmed by structured diagnostic interview (Chinese mini version) and assessment of symptom severity (Hamilton Depression Scale-17, HAMD-17) will be enrolled in a six-month open study. Healthy controls matched for age, sex and body-mass index (BMI) will have only baseline stool and electroencephalography (EEG) collections. We then will make an assessment of HAMD-17, patient-reported outcomes, and EEGs identified at the pre-treatment and those same parameters at the 1- to 6-month point. Treatment response (50% reduction in HAMD-17), treatment remission (HAMD-17<7, at least 3 weeks) will be analyzed with change in microbiome, inflammation markers and EEG.

We will analyze the differences in the intestinal flora community structure and diversity of patients and controls in order to obtain information on key different bacteria. We will conduct the correlation between each genus of bacteria in the intestinal flora and the total score of HAMD-17 in order to reveal the dynamic succession change of the intestinal flora with the disease state of major depressive disorder. The analysis with multiple testing corrections will be analyzed between depressive severity, EEG and gut microbiome composition.

The results of this study will provide the objective and direct biomarkers for major depressive disorder to achieve remission. This study will bring an important scientific basis to further optimizing treatment methods and improvie clinical effect.

ELIGIBILITY:
Inclusion Criteria:

* The proportion between male and female in each of groups was 1:1
* Han Chinese
* Permanent resident population of Beijing
* Body Mass Index,18.5-23.9
* Signed informed consent

Exclusion Criteria:

* Other severe mental disease diagnosis
* Alcohol and other substance abuse or dependence
* Patients with contraindicated signs of duloxetine
* A history of clinically significant physical disorders, including any cardiovascular, liver, kidney, respiratory, blood, endocrine, and neurological disorders, as well as clinically significant laboratory abnormalities of unstable or expected therapeutic intervention during the study period
* The apparent risk of suicide and/or the patient is considered by the investigator to be at serious risk of suicide
* Patients who had received antibiotics, probiotics and hormones within one month

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: case : 30 patients of major depressive disorder Male or female participants ages 20-40 with Major Depressive Disorder, Intervention: Drug: duloxetine control：10 subjects without major depressive disorder
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-04-10 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
the difference between the flora | pre-treatment
  The potential differences in the microbiome between depressed patients and healthy controls

SECONDARY OUTCOMES:
the dynamic succession change of the intestinal flora | 0-1-6 months
  correlation between each genus of bacteria in the intestinal flora and the total score of HAMD-17

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chao-Yang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No